CLINICAL TRIAL: NCT01866748
Title: Investigation on Safety, Tolerability and Pharmacokinetics of Single and Multiple Doses of a Long-acting GLP-1 Analogue (Semaglutide) in an Oral Formulation in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9928-4048; 2012-003199-38 (EudraCT Number); U1111-1132-4190 (Other: WHO)
Record Dates: First submitted 2013-05-22; First posted 2013-05-31 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (single dose) (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- Part B (multiple dose) (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo

INTERVENTIONS:
Drug: semaglutide — A maximum of six single-dose cohorts of oral semaglutide administered according to an ascending dose design. Starting dose 2 mg, max. dose 60 mg. Progression to next dose will be based on safety evaluation. Sequential cohorts.
  Arms: Part A (single dose)
Drug: semaglutide — Oral semaglutide administered as five multiple dose cohorts, where one of the cohorts will test a different dosing condition compared to the others. End doses from 10 mg/day to 60 mg/day. Progression to next dose will be based on safety evaluation. Semi-parallel cohorts.
  Arms: Part B (multiple dose)
Drug: placebo — In each cohort of 10, eight subjects will randomised to active treatment and two to placebo.
  Arms: Part A (single dose)
Drug: placebo — In each cohort of 24, 16 subjects will be randomised to active treatment, four to placebo and four to a enhancer-containing placebo (placebo C).
  Arms: Part B (multiple dose)

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the safety, tolerability and pharmacokinetics (the effect of the investigated drug on the body) of single and multiple doses of a long-acting GLP-1 analogue (semaglutide) in an oral formulation in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male subject, who is considered to be generally healthy, based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and laboratory safety tests performed during the screening visit, as judged by the investigator
* Body Mass Index (BMI) between 20 and 30 kg/m^2
* Glycosylated haemoglobin (HbA1c) below 6.0% (only in Part B)

Exclusion Criteria:

* History of, or presence of, cancer, diabetes or any clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal (GI), endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders, as judged by the investigator
* Use of prescription or non-prescription medicinal and herbal products (except routine vitamins) within three weeks preceding the dosing. Occasional use of paracetamol or acetylsalicylic acid is permitted

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Part A: Number of treatment emergent adverse events (TEAEs) | Day -1 to Day 24
Part B: Number of treatment emergent adverse events (TEAEs) | Recorded from the time of first dosing (Visit 3, Day -1 to day +2) and until completion of the post treatment follow-up visit (Visit 18, Day 90-104)

SECONDARY OUTCOMES:
Part A: AUC0-24h,semaglutide: the area under the semaglutide plasma concentration curve | From time 0 to 24 hours after a single dose (Day 0)
Part B: AUCτ,semaglutide: area under the semaglutide plasma concentration curve | Over the dosing interval (0-24 hours) after the last 3 daily doses (Days 67-69)
Part B: Change in fasting plasma glucose (FPG) from baseline | Day 0 (pre-dose), day 70
Part B: Change in body weight from baseline | Day -1, day 70

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Berlin, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com